CLINICAL TRIAL: NCT01095770
Title: Left Atrial Ablation With Permanent Pacemaker or ImplanTable Loop Recorder Follow-UP
Acronym: LAAPITUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Dr AN Sulke, East Sussex NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAAPITUP
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation; Atrial Fibrillation Ablation; Atrial Fibrillation monitoring; Ablation Frontiers; Reveal XT; LASSO
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ablation Frontiers Ablation (Active Comparator): This group will undergo AF ablation using Ablation Frontiers Technology.
  Interventions: Procedure: AF Ablation with Ablation Frontiers Technology
- LASSO ablation (Active Comparator): This group will undergo atrial fibrillation ablation with traditional LASSO technology
  Interventions: Procedure: AF Ablation with LASSO catheter
- Reveal XT monitoring (Active Comparator): This group will be monitored pre and post ablation using a Reveal XT implantable loop recorder.
  Interventions: Device: Reveal XT
- Permanent Pacemaker - dual chamber (Active Comparator): This group will be monitored pre and post ablation with a dual chamber permanent pacemaker
  Interventions: Device: Permanent Dual Chamber Pacemaker

INTERVENTIONS:
Procedure: AF Ablation with Ablation Frontiers Technology — AF Ablation with Ablation Frontiers Technology - PVAC, TVAC and MASC.
  Arms: Ablation Frontiers Ablation
Procedure: AF Ablation with LASSO catheter — AF Ablation with traditional LASSO catheter
  Arms: LASSO ablation
Device: Reveal XT — Reveal XT implantable loop recorder monitored group
  Arms: Reveal XT monitoring
Device: Permanent Dual Chamber Pacemaker — This group will be monitored with a dual chamber pacemaker with advanced AF monitoring capabilities.
  Arms: Permanent Pacemaker - dual chamber

SUMMARY:
The purpose of this study is 3 fold:-

1. To compare the efficacy and complication rates of 2 widely used methods, conventional irrigation tip ablation catheter (LASSO) and Ablation Frontiers ablation technology, of AF ablation for PAF.
2. To evaluate the Reveal XT ILR as a long term accurate AF monitoring device as compared to the 'gold standard' DDD pacemaker Holter.
3. To accurately evaluate, by continuous rhythm monitoring for 1 year, the efficacy of AF ablation therapy for PAF.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 16-80 years old.
* Symptomatic PAF with AF episodes self terminating after at least 30 seconds but not longer than 24 hours. Preference is given to patients with AF episodes lasting no longer than 4 hours.
* PAF should have failed at least one drug therapy medical therapy.
* Patients must give written informed consent form prior to participating in this study.

Exclusion Criteria:

* Patient is suffering with unstable angina in last 1 week.
* Patient has had a myocardial infarction within last 2 months.
* Patient is expecting or has had major cardiac surgery within last 2 months.
* Patient is participating in a conflicting study.
* Patient is mentally incapacitated and cannot consent or comply with follow-up.
* Patient has NYHA class III/ IV heart failure.
* Patients with severe valvular or ventricular dysfunction.
* Pregnancy.
* Patient suffers with other cardiac rhythm disorders.
* Recent coronary artery intervention or other factors suggesting clinical instability (ECG, clinical or laboratory findings)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
AF Burden | 12 Months
  AF Burden post left atrial ablation is defined as the sum of the duration of all atrial tachyarrhythmias expressed as a percentage of the total observation period as assessed by PM Holters.
AF Burden | 12 months
  Comparison of AF burden post PVI ablation using a conventional irrigation tip catheter with LASSO guidance (or equivalent) versus Ablation Frontiers Technology using the PVAC, MASC and TVAC catheters via standard trans-septal techniques.
AF Burden detected | 12 months
  To evaluate the Reveal XT ILR as a long term accurate AF monitoring device as compared to the 'gold standard' DDD pacemaker Holter.

SECONDARY OUTCOMES:
Arrhythmia frequency - symptomatic or asymptomatic. | 12 months
  Arrhythmia Frequency is defined as the total number of atrial tachyarrhythmic episodes divided by the observation period, expressed as episodes per day as assessed by PM Holters.
Time to first episode of AF | 12 months
  Time to persistent AF is defined as the time from ablation to the first recorded episode of AF
Average AF duration | 12 months
  Average arrhythmia duration is defined as the total duration of atrial arrhythmia divided by the total number of atrial arrhythmia episodes.
Time to persistent AF. | 12 months
  Time to persistent AF (atrial fibrillation episode lasting for 7 days)
Average SR duration. | 12 months
  Average sinus rhythm duration is defined as the total duration of sinus rhythm from first atrial arrhythmic episode until last atrial arrhythmic episode divided by the number of atrial arrhythmic episodes minus 1.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Furniss, FRCP, MD, Principal Investigator — East Sussex NHS Trust; AN Sulke, FRCP, MD, Principal Investigator — East Sussex NHS Trust
Locations (1):
- Eastbourne District General Hospital, Eastbourne, East Sussex, United Kingdom

REFERENCES:
- [Derived] Podd SJ, Sulke AN, Sugihara C, Furniss SS. Phased multipolar radiofrequency pulmonary vein isolation is as effective and safe as conventional irrigated point-to-point ablation. A prospective randomised 1-year implantable cardiac monitoring device follow-up trial. J Interv Card Electrophysiol. 2015 Dec;44(3):257-64. doi: 10.1007/s10840-015-0042-0. Epub 2015 Aug 27. PMID 26310300